CLINICAL TRIAL: NCT02024516
Title: The Effect of Concentrated Pomegranate Juice Consumption on Lipid Profile and Inflammatory Factors in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Maryam Zare, Nutritionist, Ahvaz Jundishapur University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRCT2013091614680N1
Record Dates: First submitted 2013-12-14; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Pomegranate; Inflammation; lipid profiles
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation

ARMS (1):
- 50 gr concentrated pomegranate juice (Experimental)
  Interventions: Other: 50 gr concentrated pomegranate juice

INTERVENTIONS:
Other: 50 gr concentrated pomegranate juice

SUMMARY:
The aim of this study is to examine the effects of concentrated pomegranate juice on serum lipid profile and some inflammatory factors in patients with type 2 diabetes. Forty patients aged between 25-60 years old from both sexes are recruited. Patients consume 50gr/day concentrated pomegranate juice for 4 weeks. Anthropometric and blood pressure measurements, 3-days food-record questionnaire ,physical activity and fasting blood samples were collected at the beginning and at the end of the study. Fasting blood sugar, lipid profile, TNF- a, IL-6,hs -CRP and adiponectin levels are measured. LDL are calculated by formula. The participants are asked not to change their regular diet, medicine and activity during the study.

ELIGIBILITY:
Inclusion Criteria:

* male or female 25 to 60 years old
* having type 2 diabetes for at least 6 month

Exclusion Criteria:

* pregnancy
* lactation
* cardiac disease
* hepatic disease
* respiratory disease
* chronic renal diseases
* acute or chronic inflammation
* retinopathy
* intake of antioxidant supplement
* insulin therapy
* sensitivity to concentrated pomegranate juice
* change oral drug for controlling blood glucose

Ages: 25 Years to 60 Years | Sex: All
Age Groups: Adult
Dates: Start 2013-01; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Triglyceride change | Baseline and after 4 weeks
Total Cholesterol change | Baseline and after 4 weeks
HDL- Cholesterol change | Baseline and after 4 weeks
LDL- Cholesterol change | Baseline and after 4 weeks
hsCRP change | Baseline and after 4 weeks
TNF- α change | Baseline and after 4 weeks
IL-6 change | Baseline and after 4 weeks
adiponectin change | Baseline and after 4 weeks

SECONDARY OUTCOMES:
Fasting Blood Sugar change | baseline and after 4 weeks
Blood Pressure change | Baseline and after 4 weeks
Body Mass Index change | baseline and after 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ahvaz Jundishapoor University of Medical Sciences, Ahvāz, Khoozestan, Iran